CLINICAL TRIAL: NCT05826808
Title: The Different Diagnostic Values of Polysomnographies at Low and at Moderate Altitude - A Randomized Crossover Trial
Brief Title: Effect of Moderate Altitude (>1000 m.a.s.l.) on Sleep Examinations (Polysomnography).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tsogyal Latshang (Other)
Responsible Party: Sponsor-Investigator, Tsogyal Latshang, Head of Pneumology, Kantonsspital Graubünden
Organization: Kantonsspital Graubünden (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-00636
Record Dates: First submitted 2023-03-15; First posted 2023-04-24 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): Polysomnographies will be done first for 2 nights at the sleep laboratory in Chur (600 m.a.s.l.) and after a two-week washout period for 2 nights at the participants home elevations (>1000 m.a.s.l.).
  Interventions: Diagnostic Test: Polysomnography
- B (Experimental): Polysomnographies will be done first for 2 nights at the participants home elevations (>1000 m.a.s.l.). and after a two-week washout period for 2 nights at sleep laboratory in Chur (600 m.a.s.l.).
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — The polysomnographic recordings include electroencephalogram (EEG), electrooculogram (EOG), electromyogram (EMG), electrocardiogram (ECG), pulse oximetry, transcutaneous capnography, nasal airflow and thoracic and abdominal respiratory effort.

SUMMARY:
The purpose of this study is to investigate the effect of moderate altitude (>1000 m.a.s.l.) on sleep examinations (polysomnography).

DETAILED DESCRIPTION:
Polysomnographies will be done for each participant for 2 consecutive nights at the sleep laboratory in Chur (CH; 600 m.a.s.l.) as well as for 2 consecutive nights at the participants home elevations (CH; >1000 m.a.s.l.). Between the measurements at those two different altitudes there will be a two-week washout period at >1000 m.a.s.l.. The sequence of altitude exposure will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no current medical condition or intake of regular medication, except negligible medical issues or accidents not interfering with the current health status or physical performance.)
* Living above 1000 m.a.s.l. since at least 1 year
* No overnight stay at altitudes <1000 m.a.s.l. in the previous 4 weeks
* 18-70 years old
* Body mass index 18,5-30 kg/m2
* informed consent

Exclusion Criteria:

* Active diseases or health related conditions that require treatment (sleep disorders (mainly sleep apnea), chronic rhinitis, cardiovascular and lung diseases)
* Use of drugs that affect the respiratory center drive (sedatives, sleep inducing drugs, opioids), stimulants or illegal drugs
* Regular consumption of recreational drugs (alcohol and nicotine included)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
T90 (time spent in SpO2 below 90%) | 4 nights
  T90 is the percent of sleeping time which the participant spent in SpO2 below 90%. It provides information about the duration and degree of hypoxia during the whole sleep.

SECONDARY OUTCOMES:
SpO2 (oxygen saturation) | 4 nights
  SpO2 is the amount of haemoglobin bound to oxygen. Normal values lie above 95%. Values below 90% are considered as low and require treatment.
AHI (apnea-hypopnea index) | 4 nights
  AHI is defined as the number of apneas and hypopneas per hour of sleep, whereby apnea is defined as a cessation of the airflow for ≥10 seconds, while hypopnea is defined as a reduction of the airflow ≥30% with an oxygen desaturation ≥3% or an arousal.
SWS (slow-wave sleep) | 4 nights
  SWS includes the deep sleep phase. Deep sleep is amongst other important for energy restoration, immune system strengthening and regeneration of cells.
AI (arousal index) | 4 nights
  AI is the number of arousals per hour of sleep, whereby an arousal is an interruption of sleep from 3-15 seconds. They prevent suffocation in the sleep apnea by interrupting breathing pauses but are also coupled with a lot of stress for the human body.
TcCO2 (partial pressure of carbon dioxide) | 4 nights
  TcCO2 correlates with PaCO2 and is therefore a non-invasive alternative. A normal value of PCO2 lies between 35 and 45 mmHg. Lower values can lead to muscle cramps, abnormal heartbeat and much more.
WASO (wakefulness after sleep onset) | 4 nights
  WASO is the time spent awake after sleep onset. High values of WASO are for example found in sleep apnea, insomnia and restless leg syndrome.
ODI (oxygen desaturation index) | 4 nights
  ODI is defined as the number of oxygen decreases ≥3% per hour of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Tsogyal Latshang, PD Dr. med., Principal Investigator — Kantonsspital Graubünden
Locations (1):
- Kantonsspital Graubünden, Chur, Switzerland

IPD SHARING:
Plan to Share IPD: No